CLINICAL TRIAL: NCT01231503
Title: Safety and Immunogenicity of GSK Biologicals' Candidate Malaria Vaccine 257049 When Administered on Different Schedules to Infants in Africa
Brief Title: Safety and Immunogenicity of GSK Biologicals' Malaria Vaccine 257049 When Administered on 7 Schedules to African Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111315
Record Dates: First submitted 2010-10-14; First posted 2010-11-01 (Estimated); Results first posted 2015-05-20 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-06

CONDITIONS: Malaria
Keywords: Africa; malaria vaccine; schedule; EPI; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Engerix-B; Measles Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- RTS,S Neo-10-14 Group (Experimental): Subjects received 3 doses of RTS,S/AS01E (GSK257049) when ≤ 7 days of age and at 10 and 14 weeks of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when ≤7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- RTS,S Neo-10-26 Group (Experimental): Subjects received 3 doses of RTS,S/AS01E (GSK257049) when ≤ 7 days of age and at 10 and 26 weeks of age. In addition, all subjects received a 3-doses course of Tritanri xHepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when below ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- RTS,S 6-10-14 Group (Experimental): Subjects received 3 doses of RTS,S/AS01E (GSK257049) at 6, 10 and 14 weeks of age In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- RTS,S 6-10-26 Group (Experimental): Subjects received 3 doses of RTS,S/AS01E (GSK257049) at 6, 10 and 26 weeks of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- Engerix-B Neo/RTS,S 6-10-26 Group (Experimental): Subjects received one dose of Engerix-B (HBV) when ≤ 7 days of age followed by 3 doses of RTS,S/AS01E (GSK257049) at 6, 10 and 26 weeks of age In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E and HBV vaccines were administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Engerix-B; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- RTS,S 10-14-26 Group (Experimental): Subjects received 3 doses of RTS,S/AS01E (GSK257049) at 10, 14 and 26 weeks of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when below ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- RTS,S 14-26-9M Group (Experimental): Subjects received 3 doses of RTS,S/AS01E (or GSK257049) at 14 and 26 weeks of age and at 9 months of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when below ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when below ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: GSK Biological's Investigational Malaria Vaccine 257049; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax
- Engerix-B Neo Group (Active Comparator): Subjects in this group received one dose of Engerix-B (HBV) ≤ 7 days of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when below ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The HBV vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
  Interventions: Biological: Engerix-B; Biological: Tritanrix HepB Hib; Biological: BCG; Biological: OPV; Biological: Rouvax

INTERVENTIONS:
Biological: GSK Biological's Investigational Malaria Vaccine 257049 — 3 doses, intramuscular (IM) route, in left antero-lateral thigh, as follows: 1) RTS,S Neo-10-14 Group at less than (=<) 7 days, at 10 and 14 weeks (wks) of age; 2) RTS,S Neo-10-26 Group =< 7 days, at 10 and 26 wks of age; 3) RTS,S 6-10-14 Group at 6, 10 and 14 wks of age; 4) RTS,S 6-10-26 Group at 6, 10 and 26 wks of age; 5) Engerix-B Neo/RTS,S 6-10-26 Group at 6, 10 and 26 wks of age; 6) RTS,S 10-14-26 Group at 10, 14 and 26 wks of age; 7) RTS,S 14-26-9M Group at 14 and 26 wks of age and at 9 months of age
  Other Names: GSK257049; RTS; S/AS01E
  Arms: Engerix-B Neo/RTS,S 6-10-26 Group; RTS,S 10-14-26 Group; RTS,S 14-26-9M Group; RTS,S 6-10-14 Group; RTS,S 6-10-26 Group; RTS,S Neo-10-14 Group; RTS,S Neo-10-26 Group
Biological: Engerix-B — 1 dose, intramuscular route: left antero-lateral thigh at birth (=< 7 days of age)
  Other Names: HBV
  Arms: Engerix-B Neo Group; Engerix-B Neo/RTS,S 6-10-26 Group
Biological: Tritanrix HepB Hib — 3 doses, intramuscular route: right antero-lateral thigh at 6, 10 and 14 weeks of age
  Other Names: DTPwHepB/Hib
Biological: BCG — 1 dose, intradermal route, in shoulder at birth (=< 7 days of age)
  Other Names: Bacille Calmette Guerin tuberculosis vaccine
Biological: OPV — 4 doses, orally, at birth (=< 7 days of age) and at 6, 10 and 14 weeks of age
  Other Names: Polio Sabin
Biological: Rouvax — 1 dose, intramuscular (IM) route, in left antero-lateral thigh, at 9 months of age
  Other Names: Measles; measles vaccine

SUMMARY:
The aim of the malaria vaccine program of the MVI/GSK partnership is to develop an efficacious malaria vaccine that is deliverable through the existing system, the Expanded Program on Immunization (EPI) of WHO. This study has been designed to:

* Investigate the safety and immunogenicity of 7 infant immunization schedules of the experimental malaria vaccine integrated with an EPI regimen.
* Investigate how to maximize the antibody response to the experimental malaria vaccine.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* A male or female infant between 1 and 7 days (inclusive) of age (where day 1 is day of birth).
* Signed or thumb-printed informed consent obtained from the parent(s)/guardian(s) of the child. Where parent(s)/guardian(s) are illiterate, the consent form will be countersigned by a witness.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. return for follow-up visits) should be enrolled in the study.
* Born to a mother negative for HIV antibody and Hepatitis B surface antigen.
* Subjects who are born after a normal gestation period (between 37 and 42 weeks) (Gestational age will be determined by carrying out a clinical assessment on infants according to the principles set out by Dubowitz (1970) in the first 5 days of life).
* A minimum weight of 2.5 kg.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* Acute or chronic illness determined by clinical or physical examination and laboratory screening tests including, but not limited to:

  * Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
  * A family history of congenital or hereditary immunodeficiency.
  * Major congenital defects.
  * History of any neurological disorders or seizures.
* Laboratory screening tests out of normal ranges/limits defined per protocol.
* Previous vaccination with diphtheria, tetanus, pertussis (whole-cell or acellular), Hemophilus influenzae type b, hepatitis B, BCG tuberculosis, measles or oral polio vaccines.
* Planned administration/administration of a licensed vaccine (i.e. a vaccine that is approved by one of the following authorities: FDA or EU member state or WHO [with respect to prequalification]) not foreseen by the study protocol within 7 days of the first dose of study vaccine.
* Administration of immunoglobulins, blood transfusions or other blood products since birth to the first dose of study vaccine or planned administration during the study period.
* Use of a drug or vaccine that is not approved for that indication (by one of the following authorities: FDA or EU member state or WHO [with respect to prequalification]) other than the study vaccine starting at birth or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Simultaneous participation in any other clinical trial.
* Same-sex twins (to avoid misidentification).
* Maternal death.
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Children will not be enrolled if any maternal, obstetrical or neonatal event that has occurred might, in the judgment of the investigator, result in increased neonatal/infant morbidity
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Actual)
Dates: Start 2011-01-13 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangwe, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Witte D, Cunliffe NA, Turner AM, Ngulube E, Ofori-Anyinam O, Vekemans J, Chimpeni P, Lievens M, Wilson TP, Njiram'madzi J, Mendoza YG, Leach A. Safety and Immunogenicity of Seven Dosing Regimens of the Candidate RTS,S/AS01E Malaria Vaccine Integrated Within an Expanded Program on Immunization Regimen: A Phase II, Single-Center, Open, Controlled Trial in Infants in Malawi. Pediatr Infect Dis J. 2018 May;37(5):483-491. doi: 10.1097/INF.0000000000001937. PMID 29432383
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 480 subjects were enrolled into the study. Out of these 480 subjects, 479 were vaccinated and 1 was allocated a subject number but was not vaccinated.
Pre-assignment Details: 480 subjects were enrolled into the study. Out of these 480 subjects, 479 were vaccinated and 1 was allocated a subject number but was not vaccinated.
Groups:
- RTS,S Neo-10-26 Group: Subjects received 3 doses of RTS,S/AS01E (GSK257049) when ≤ 7 days of age and at 10 and 26 weeks of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when below ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
Period: Overall Study
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Started | 60 | 59 | 60 | 60 | 60 | 60 | 60 | 60
Completed | 46 | 46 | 48 | 52 | 50 | 44 | 53 | 52
Not Completed | 14 | 13 | 12 | 8 | 10 | 16 | 7 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse event, serious fatal | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 3 | 3 | 1 | 3 | 5 | 1 | 2
Not completed — Lost to Follow-up | 8 | 10 | 8 | 5 | 7 | 9 | 6 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RTS,S 10-14-26 Group: Subjects received 3 doses of RTS,S/AS01E (GSK257049) at 10, 14 and 26 weeks of age. In addition, all subjects received a 3-doses course of TritanrixHepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when below ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
- Total: Total of all reporting groups
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group | Total
Number analyzed (Participants) | 60 | 59 | 60 | 60 | 60 | 60 | 60 | 60 | 479
Age, Continuous [Mean (Standard Deviation); unit: Days] | 0.4 (1.1) | 0.4 (1.2) | 0.2 (1.0) | 0.2 (0.8) | 0.5 (1.4) | 0.2 (0.8) | 0.2 (0.9) | 0.4 (1.2) | 0.3 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 28 | 35 | 31 | 29 | 24 | 28 | 237
  Male | 30 | 27 | 32 | 25 | 29 | 31 | 36 | 32 | 242

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reported With Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or may evolve into one of the outcomes listed above. "Any" is defined an incidence of a SAE regardless of intensity/severity.
Time Frame: From study start at Month 0 up to Month 10.
Population: Analysis was done on the Total Vaccinated cohort, which included all subjects who were randomized and received a dose of BCG tuberculosis vaccine. Analyses on this cohort were performed per treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 60 | 59 | 60 | 60 | 60 | 60 | 60 | 60
Participants | 5 | 4 | 5 | 7 | 5 | 10 | 4 | 3

2. Primary Outcome: Concentrations of Antibodies Against Circumsporozoite Protein of Plasmodium Falciparum (Anti-CS Antibodies)
Description: Anti-CS antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs) expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off for the endpoint was a GMC value greater than or equal to (≥) 0.5 EL.U/mL.
Time Frame: At 1 month (M) post Dose 3 of RTS,S/AS01E, e. a. M5 for RTS,S Neo-10-14, RTS,S 6-10-14 and Engerix-B Neo groups
Population: Analysis was done on the According-to-Protocol cohort for immunogenicity, that is, subjects from the Total Vaccinated cohort who received all vaccinations, complied to protocol procedures, and for whom results were available for the antibody concentrations/titers assessed in the specified outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S 6-10-14 Group | Engerix-B Neo Group
Number analyzed (Participants) | 47 | 45 | 48
EL.U/mL | 128.2 [92.2 to 178.2] | 218.3 [160.1 to 297.6] | 0 [0 to 0]

3. Primary Outcome: Concentrations of Antibodies Against Circumsporozoite Protein of Plasmodium Falciparum (Anti-CS Antibodies)
Description: as for outcome 2
Time Frame: At 1 month (M) post Dose 3 of RTS,S/AS01E, e. a. M7 for RTS,S Neo-10-26, RTS,S 6-10-26, Engerix-B Neo/RTS,S 6-10-26, and RTS,S 10-14-26 groups
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Neo-10-26 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group
Number analyzed (Participants) | 43 | 46 | 43 | 41
EL.U/mL | 136.6 [93 to 200.7] | 156.5 [100.4 to 244] | 170.6 [114.6 to 254.1] | 392.6 [323.3 to 476.7]

4. Primary Outcome: Concentrations of Antibodies Against Circumsporozoite Protein of Plasmodium Falciparum (Anti-CS Antibodies)
Description: as for outcome 2
Time Frame: At 1 month (M) post Dose 3 of RTS,S/AS01E, e. a. M10 for RTS,S 14-26-9M Group
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S 14-26-9M Group
Number analyzed (Participants) | 47
EL.U/mL | 269.9 [183.3 to 397.5]

5. Secondary Outcome: Number of Subjects Reported With Unsolicited Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. "Any" is defined an incidence of an unsolicited AE regardless of intensity or relationship to study vaccination. Please note that, for this outcome measure, analysis was performed only on subjects with at least one administered dose of RTS,S/AS01E and/or DTPwHepB/Hib for the Engerix-B Neo Group.
Time Frame: During the 30-day (Days 0-29) post vaccination period following 3 doses of RTS,S/AS01E versus DTPwHepB/Hib for the Engerix-B Neo Group
Population: Analysis was done on the Total Vaccinated cohort, which included all subjects who were randomized and received a dose of BCG tuberculosis vaccine. Analyses on this cohort were performed per treatment assignment. This analysis was done solely on subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 60 | 59 | 54 | 57 | 57 | 52 | 57 | 52
Participants | 36 | 35 | 28 | 29 | 35 | 36 | 47 | 31

6. Secondary Outcome: Number of Subjects Reported With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From study start at Month 0 up to Month 18 (corresponding data lock point =23 March 2015)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 60 | 59 | 60 | 60 | 60 | 60 | 60 | 60
Participants | 7 | 5 | 6 | 9 | 8 | 12 | 5 | 4

7. Secondary Outcome: Number of Subjects Reported With Biochemical Abnormalities, for the Alanine Aminotransferase (ALT) Parameter
Description: This outcome measure concerns biochemical abnormalities, for the alanine aminotransferase (ALT) parameter. Subjects' levels were assessed as either normal, Grade 1, Grade 2, Grade 3, Grade 4 or Missing. Normal ALT level was defined as ALT< 60 International units per milliliter (IU/mL). Grade 1 ALT level was defined as 1.1 to 2.5 times the upper limit of normal (ULN). Grade 2 ALT level was defined as 2.6 to 5.0 times the ULN. Grade 3 ALT level was defined as 5.1 to 10.0 times the ULN. Grade 4 ALT level was defined as > 10.0 times the ULN.
Time Frame: At Day 7 post dose 1 (7D+W6) and at Day 30 post dose 3 (30D+W14).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 58 | 57 | 53 | 57 | 57 | 54 | 57 | 58
Participants
  7D+W6, Normal | 56 | 55 | 51 | 55 | 55 | 52 | 56 | 57
  7D+W6, Grade 1 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1
  7D+W6, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Missing | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0
  30D+W14, Normal: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Normal | 48 | 49 | 49 | 52 | 52 | 47 | 51 | 50
  30D+W14, Grade 1: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 2: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 3: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 4: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Missing: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Missing | 2 | 0 | 1 | 2 | 1 | 0 | 2 | 1

8. Secondary Outcome: Number of Subjects Reported With Biochemical Abnormalities, for the Creatinine (CREA) Parameter
Description: This outcome measure concerns biochemical abnormalities, for the creatinine (CREA) parameter. Subjects' levels were assessed as either normal, Grade 1, Grade 2, Grade 3, Grade 4 or Missing. Normal CREA level was defined as CREA ≤ 106, 88 and 71 micromoles per liter (µmol/L) for subjects 1, 2 or ≥ 2 days of age, respectively. Grade 1 CREA level was defined as 1.1 to 1.3 times the upper limit of normal (ULN). Grade 2 CREA level was defined as 1.4 to 1.8 times the ULN. Grade 3 CREA level was defined as 1.9 to 3.4 times the ULN. Grade 4 CREA level was defined as ≥ 3.5 times the ULN.
Time Frame: At Day 7 post dose 1 (7D+W6) and at Day 30 post dose 3 (30D+W14).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 58 | 57 | 53 | 57 | 57 | 54 | 57 | 58
Participants
  7D+W6, Normal | 55 | 55 | 53 | 57 | 57 | 53 | 57 | 56
  7D+W6, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Missing | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 2
  30D+W14, Normal: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Normal | 50 | 49 | 50 | 52 | 53 | 47 | 51 | 50
  30D+W14, Grade 1: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 2: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 3: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 4: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Missing: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 53 | 51
  30D+W14, Missing | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1

9. Secondary Outcome: Number of Subjects Reported With Haematological Abnormalities, for the Haemoglobin (HAE) Parameter
Description: This outcome measure concerns haematological abnormalities, for the haemoglobin (HAE) parameter. Subjects' levels were assessed as either normal, Grade (G) 1, G 2, G 3, G 4 or Missing. Normal HAE level was defined as HAE > 13.0 and 10.5 grams per deciliter (g/dL) for subjects aged 1 to 21 and 22 to 35 days respectively. Grades were defined as follows: 1) In subjects aged 1 to 21 days: G1 = HAE as 12.0 to 13.0 g/dL, G2 = HAE as 10.0 to 11.9 g/dL, G3 = HAE as 9.0 to 9.9 g/dL, G4 = HAE < 9.0 g/dL; 2) In subjects aged 22 to 35 days: G1 = HAE as 9.5 to 10.5 g/dL, G2 = HAE as 8.0 to 9.4 g/dL, G3 = HAE as 7.0 to 7.9 g/dL, G4 = HAE < 7.0 g/dL; 3) In subjects aged 36 to 56 days: G1 = HAE as 8.5 to 9.4 g/dL, G2 = HAE as 7.0 to 8.4 g/dL, G3 = HAE as 6.0 to 6.9 g/dL, G4 = HAE < 6.0 g/dL; 4) In subjects aged ≥ 57 days: G1 = HAE as 10.0 to 10.9 g/dL, G2 = HAE as 9.0 to 9.9 g/dL, G3 = HAE as 7.0 to 8.9 g/dL, G4 = HAE < 7.0 g/dL.
Time Frame: At Day 7 post dose 1 (7D+W6) and at Day 30 post dose 3 (30D+W14).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 58 | 57 | 53 | 57 | 57 | 54 | 57 | 58
Participants
  7D+W6, Grade 1 | 1 | 5 | 5 | 5 | 7 | 6 | 21 | 3
  7D+W6, Grade 2 | 5 | 4 | 2 | 0 | 2 | 2 | 9 | 3
  7D+W6, Grade 3 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 3
  7D+W6, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  7D+W6, Missing | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  30D+W14, Normal: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Normal | 25 | 17 | 23 | 15 | 12 | 6 | 15 | 20
  30D+W14, Grade 1: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 1 | 16 | 15 | 16 | 18 | 26 | 15 | 19 | 24
  30D+W14, Grade 2: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 2 | 7 | 11 | 10 | 13 | 11 | 18 | 12 | 6
  30D+W14, Grade 3: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 3 | 3 | 6 | 0 | 7 | 4 | 8 | 8 | 2
  30D+W14, Grade 4: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  30D+W14, Missing: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  7D+W6, Normal | 51 | 47 | 43 | 50 | 48 | 45 | 25 | 48

10. Secondary Outcome: Number of Subjects Reported With Haematological Abnormalities, for the Platelets (PLA) Parameter
Description: This outcome measure concerns haematological abnormalities, for the platelets (PLA) parameter. Subjects' levels were assessed as either normal, Grade (G) 1, G2, G3, G4 or Missing. Normal PLA level was defined as > 125 x 10 exp 9 PLA per liter (Billions PLA/L). Grade 1 PLA level was defined as 100 to 125 Billions PLA/L. Grade 2 PLA level was defined as 50 to 99 Billions PLA/L. Grade 3 PLA level was defined as 25 to 49 Billions PLA/L. Grade 4 PLA level was defined as < 25 Billions PLA/L.
Time Frame: At Day 7 post dose 1 (7D+W6) and at Day 30 post dose 3 (30D+W14).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 58 | 57 | 53 | 57 | 57 | 54 | 57 | 58
Participants
  7D+W6, Grade 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 5
  7D+W6, Grade 2 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 2
  7D+W6, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Missing | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0
  30D+W14, Normal: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Normal | 51 | 49 | 46 | 53 | 51 | 45 | 53 | 51
  30D+W14, Grade 1: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0
  30D+W14, Grade 2: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  30D+W14, Grade 3: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 4: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 4 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  30D+W14, Missing: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  7D+W6, Normal | 54 | 55 | 47 | 55 | 57 | 53 | 57 | 51

11. Secondary Outcome: Number of Subjects Reported With Haematological Abnormalities, for the White Blood Cells (WBC) Parameter
Description: This outcome measure concerns haematological abnormalities, for the white blood cells (WBC) parameter. Subjects' levels were assessed as either normal, Grade 1, Grade 2, Grade 3, Grade 4 or Missing. Normal WBC level was defined as > 2.5 x 10 exp 9 WBC per liter (Billions WBC/L). Grade 1 WBC level was defined as 2.0 to 2.5 Billions WBC/L. Grade 2 WBC level was defined as 1.5 to 1.999 Billions WBC/L. Grade 3 WBC level was defined as 1.0 to 1.499 Billions WBC/L. Grade 4 WBC level was defined as < 1.0 Billions WBC/L.
Time Frame: At Day 7 post dose 1 (7D+W6) and at Day 30 post dose 3 (30D+W14).
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 58 | 57 | 53 | 57 | 57 | 54 | 57 | 58
Participants
  7D+W6, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  7D+W6, Missing | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
  30D+W14, Normal: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Normal | 51 | 49 | 50 | 53 | 53 | 47 | 54 | 52
  30D+W14, Grade 1: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 2: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 3: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Grade 4: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  30D+W14, Missing: number analyzed (Participants) | 51 | 49 | 50 | 54 | 53 | 47 | 54 | 52
  30D+W14, Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  7D+W6, Normal | 57 | 57 | 50 | 56 | 57 | 54 | 57 | 58

12. Secondary Outcome: Concentrations of Antibodies Against Circumsporozoite Protein of Plasmodium Falciparum (Anti-CS Antibodies)
Description: Anti-CS antibody concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean concentrations (GMCs) expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off value for the assay was greater than or equal to (≥) 0.5 EL.U/mL.
Time Frame: At Screening (SCR), at Month (M) 4, at M5, at M7 and/or at M10, according to the vaccination scheduling for the specific group assessed concerned group
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 47 | 43 | 45 | 46 | 45 | 44 | 51 | 48
EL.U/mL
  Anti-CS, at SCR: number analyzed (Participants) | 43 | 42 | 45 | 43 | 45 | 42 | 51 | 45
  Anti-CS, at SCR | 0.5 [0.4 to 0.7] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.6] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.5] | 0.5 [0.4 to 0.7]
  Anti-CS, at M4: number analyzed (Participants) | 30 | 32 | 31 | 37 | 39 | 0 | 0 | 36
  Anti-CS, at M4 | 33.6 [18.5 to 61.3] | 72.8 [44.6 to 118.7] | 112.2 [76.0 to 165.8] | 99.7 [61.3 to 162.0] | 88.0 [55.4 to 139.8] |  |  | 0 [0 to 0]
  Anti-CS, at M5: number analyzed (Participants) | 47 | 0 | 45 | 0 | 0 | 44 | 0 | 48
  Anti-CS, at M5 | 128.2 [92.2 to 178.2] |  | 218.3 [160.1 to 297.6] |  |  | 167.6 [133.2 to 210.9] |  | 0 [0 to 0]
  Anti-CS, at M7: number analyzed (Participants) | 0 | 43 | 0 | 46 | 43 | 41 | 36 | 47
  Anti-CS, at M7 |  | 136.6 [93.0 to 200.7] |  | 156.5 [100.4 to 244.0] | 170.6 [114.6 to 254.1] | 392.6 [323.3 to 476.7] | 141.7 [97.0 to 207.1] | 0 [0 to 0]
  Anti-CS, at M10: number analyzed (Participants) | 39 | 37 | 36 | 40 | 39 | 38 | 47 | 40
  Anti-CS, at M10 | 13.8 [8.5 to 22.6] | 39.5 [22.4 to 69.6] | 30.1 [18.8 to 48.2] | 44.2 [23.8 to 82.2] | 43.3 [24.6 to 76.0] | 121.0 [89.4 to 163.7] | 269.9 [183.3 to 397.5] | 0.3 [0.2 to 0.4]

13. Secondary Outcome: Anti-Hepatitis B Surface Antibody (Anti-HBs) Concentrations.
Description: Concentrations, by enzyme-linked immunosorbent assay (ELISA), were presented as geometric mean concentrations (GMCs), and expressed in milli-international units per milliliter (mIU/mL). The seropositivity and seroprotection cut-off values for the assay were greater than or equal to (≥) 6.2 and 10 mIU/mL, respectively.
Time Frame: At Screening (SCR), at Month 5 (M5), at Month 7 (M7) and at Month 10 (M10), according to the vaccination scheduling
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 33 | 37 | 37 | 38 | 37 | 34 | 37 | 38
mIU/mL
  SCR: number analyzed (Participants) | 27 | 25 | 32 | 34 | 32 | 32 | 37 | 31
  SCR | 10.7 [4.2 to 27.3] | 22.2 [6.6 to 74.6] | 9.9 [4.4 to 22.0] | 9.5 [4.4 to 20.6] | 17.2 [7.1 to 41.8] | 12.6 [4.9 to 32.0] | 38.6 [13.6 to 109.5] | 22.6 [8.5 to 59.8]
  M5: number analyzed (Participants) | 25 | 0 | 17 | 0 | 0 | 0 | 0 | 22
  M5 | 6479.0 [3858.9 to 10878.2] |  | 3831.6 [1783.4 to 8232.3] |  |  |  |  | 640.7 [381.3 to 1076.7]
  M7: number analyzed (Participants) | 0 | 35 | 0 | 37 | 30 | 34 | 0 | 38
  M7 |  | 23218.5 [16670.1 to 32339.2] |  | 29839.9 [20731.1 to 42951.0] | 34589.1 [21299.2 to 56171.6] | 44472.4 [31305.5 to 63177.1] |  | 430.1 [277.8 to 666.0]
  M10: number analyzed (Participants) | 33 | 37 | 37 | 38 | 37 | 31 | 37 | 34
  M10 | 2949.5 [2040.5 to 4263.4] | 9630.8 [6472.2 to 14330.9] | 3135.0 [2287.6 to 4296.2] | 8581.8 [5974.8 to 12326.5] | 12084.3 [8211.6 to 17783.5] | 13360.1 [8195.5 to 21779.4] | 75018.0 [54992.1 to 102336.5] | 139.5 [77.2 to 252.1]

14. Secondary Outcome: Anti-diphtheria (Anti-D) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: Anti-D and anti-TT antibody concentrations were calculated, expressed as geometric mean concentrations (GMCs), in International units per milliliter (IU/mL), and tabulated. The seropositivity cut-off value for the assay was ≥ 0.1 IU/mL.
Time Frame: At Month 5
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 48 | 46 | 45 | 48 | 47 | 44 | 54 | 47
IU/mL
  Anti-D | 3.1 [2.2 to 4.5] | 3.9 [2.9 to 5.3] | 3.2 [2.5 to 4.0] | 4.0 [3.2 to 5.1] | 3.6 [2.7 to 4.8] | 4.3 [3.2 to 5.8] | 4.3 [3.4 to 5.5] | 4.6 [3.7 to 5.6]
  Anti-TT | 3.5 [2.6 to 4.6] | 3.2 [2.3 to 4.4] | 3.7 [2.8 to 4.8] | 2.8 [2.2 to 3.7] | 3.3 [2.4 to 4.4] | 3.3 [2.4 to 4.6] | 3.5 [2.6 to 4.6] | 4.6 [3.5 to 6.0]

15. Secondary Outcome: Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: Anti-PRP antibody concentrations were calculated, expressed as geometric mean concentrations (GMCs), in microgram per milliliter (µg/mL), and tabulated. The seroprotection cut-off value for the assay was ≥ 0.15 µg/mL.
Time Frame: At Month 5
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 47 | 44 | 44 | 48 | 47 | 43 | 52 | 47
µg/mL | 6.8 [4.5 to 10.3] | 11.1 [7.5 to 16.5] | 11.4 [7.3 to 17.8] | 13.6 [9.6 to 19.3] | 10.9 [7.4 to 16.0] | 11.0 [7.1 to 16.9] | 15.6 [10.6 to 22.8] | 13.8 [9.7 to 19.5]

16. Secondary Outcome: Anti-polio Type 1, 2 and 3 (Anti-Polio 1, 2 and 3) Antibody Concentrations
Description: Anti-Polio 1, 2 and 3 antibody concentrations were calculated, expressed as geometric mean concentrations (GMCs), in international units per mililiter (IU/mL) and tabulated. The seroprotection cut-off value for the assay was ≥ 8 IU/mL.
Time Frame: At Month 5
Population: Analysis was done on the According-to-Protocol cohort for immunogenicity included all subjects included in the Total Vaccinated cohort who received all vaccinations according to protocol procedures within specified intervals and did not take any immune modifying medication or had blood transfusions.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 31 | 16 | 25 | 25 | 19 | 29 | 25 | 30
IU/mL
  Anti-Polio 1: number analyzed (Participants) | 25 | 13 | 20 | 14 | 13 | 20 | 20 | 19
  Anti-Polio 1 | 27.6 [16.5 to 46] | 21.6 [10.3 to 45.2] | 31.7 [17.2 to 58.7] | 47.1 [21.5 to 102.8] | 19.9 [4 to 98.3] | 23.6 [8.4 to 66.5] | 16.7 [7.9 to 35.4] | 45.4 [18.9 to 109.4]
  Anti-Polio 2 | 27.5 [16.8 to 45.1] | 35.1 [14.9 to 82.4] | 56.6 [32.8 to 97.7] | 37.9 [17 to 84.6] | 42 [21.6 to 81.6] | 27.6 [12.6 to 60.4] | 40.1 [24.1 to 66.6] | 25.9 [16.4 to 40.7]
  Anti-Polio 3: number analyzed (Participants) | 27 | 11 | 23 | 18 | 16 | 24 | 24 | 26
  Anti-Polio 3 | 3.6 [1.6 to 7.9] | 2.3 [0.6 to 8.7] | 5.1 [2.6 to 10.2] | 3.3 [1.3 to 8.4] | 5.6 [2.6 to 12.2] | 2.6 [1.2 to 5.7] | 3 [1.6 to 5.5] | 6 [3.3 to 10.8]

17. Secondary Outcome: Concentrations of Antibodies Against Acellular B-pertussis (BPT)
Description: Concentrations of anti-BPT antibodies were determined by enzyme-linked immunosorbent assay (ELISA) and expressed as geometric mean concentrations (GMCs), in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off value for the assay was ≥ 15 EL.U/mL.
Time Frame: At Month 5
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 43 | 42 | 41 | 46 | 42 | 42 | 50 | 41
EL.U/mL | 82.9 [69.9 to 98.4] | 102.3 [84.9 to 123.4] | 86.7 [72.5 to 103.7] | 81.2 [66.7 to 98.8] | 99.2 [82.6 to 119.1] | 86.1 [71.7 to 103.4] | 91.0 [75.9 to 109.0] | 109.8 [89.7 to 134.4]

18. Secondary Outcome: Concentrations of Antibodies Against Measles Antigens
Description: Concentrations of anti measles antibodies were determined by ELISA and expressed as GMCs in milli-international units per millilitre (mIU/mL).
  The seropositivity cut-off value for the assay was ≥ 150 mIU/mL. Please note that this outcome measure was only assessed in subjects in the RTS,S 14-26-9M and Engerix-B Neo groups.
Time Frame: At Month 10
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 52 | 46
mIU/mL | 1017.7 [751.9 to 1377.4] | 1430.6 [996.9 to 2053.2]

19. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. "Any" about a specific symptom is defined as incidence of this symptom, regardless of its intensity.
Time Frame: Within 7 days (Days 0-6) after Week 0 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 60 | 59 | 58 | 60 | 60 | 59 | 60 | 59
Participants
  Any Pain | 1 | 4 | 2 | 2 | 2 | 0 | 2 | 1
  Any Redness | 3 | 4 | 5 | 6 | 7 | 4 | 11 | 6
  Any Swelling | 2 | 4 | 5 | 6 | 5 | 5 | 8 | 6

20. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: as for outcome 19
Time Frame: Within 7 days (Days 0-6) after Week 6 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 55 | 55 | 54 | 57 | 57 | 55 | 58 | 51
Participants
  Any Pain | 2 | 2 | 7 | 7 | 3 | 6 | 4 | 6
  Any Redness | 3 | 2 | 6 | 4 | 4 | 5 | 4 | 4
  Any Swelling | 4 | 3 | 6 | 8 | 6 | 6 | 6 | 6

21. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: as for outcome 19
Time Frame: Within 7 days (Days 0-6) after Week 10 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- RTS,S 10-14-26 Group; RTS,S 14-26-9M Group: Subjects received 3 doses of RTS,S/AS01E (or GSK257049) at 14 and 26 weeks of age and at 9 months of age. In addition, all subjects received a 3-doses course of Tritanrix HepB/Hib (DTPwHepB/Hib), administered at 6, 10 and 14 weeks of age, one dose of Bacille Calmette Guerin tuberculosis vaccine (BCG), administered when below ≤ 7 days of age, 4 doses of Polio Sabin (OPV), administered when below ≤ 7 days of age and at 6, 10 and 14 weeks of age, and one dose of Rouvax (Measles), administered at 9 months of age. The RTS,S/AS01E vaccine was administered intramuscularly (IM) in the left antero-lateral thigh. The DTPwHepB/Hib and Measles vaccines were administered IM in the right antero-lateral thigh and the OPV vaccine orally. The BCG vaccine was administered via intradermal route in the shoulder.
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 52 | 54 | 51 | 54 | 56 | 52 | 57 | 51
Participants
  Any Pain | 4 | 2 | 0 | 5 | 1 | 2 | 5 | 3
  Any Redness | 2 | 1 | 1 | 4 | 2 | 3 | 6 | 3
  Any Swelling | 4 | 1 | 3 | 6 | 3 | 3 | 6 | 3

22. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: as for outcome 19
Time Frame: Within 7 days (Days 0-6) after Week 14 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 51 | 53 | 51 | 54 | 55 | 50 | 57 | 52
Participants
  Any Pain | 4 | 5 | 4 | 1 | 4 | 3 | 1 | 3
  Any Redness | 4 | 5 | 4 | 1 | 3 | 2 | 2 | 3
  Any Swelling | 7 | 5 | 4 | 1 | 4 | 4 | 2 | 3

23. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. "Any" about a specific symptom is defined as incidence of this symptom, regardless of its intensity. RTS,S Neo-10-14 Group, RTS,S 6-10-14 Group and Engerix-B Neo Group didn't receive vaccination at this time point.
Time Frame: Within 7 days (Days 0-6) after Week 26 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-26 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group
Number analyzed (Participants) | 49 | 54 | 54 | 46 | 56
Participants
  Any Pain | 0 | 0 | 0 | 0 | 0
  Any Redness | 0 | 0 | 0 | 0 | 0
  Any Swelling | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects Reported With Solicited Local Symptoms
Description: as for outcome 19
Time Frame: Within 7 days (Days 0-6) after Month 9 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 50 | 49 | 48 | 54 | 51 | 47 | 56 | 51
Participants
  Any Pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: Solicited general symptoms assessed include Drowsiness, Fever (temperature by axillary route ≥ 37.5°C), Irritability/Fussiness and Loss of appetite. "Any" about a specific symptom is defined as incidence of this symptom, regardless of its intensity or relationship to vaccination.
Time Frame: Within 7 days (Days 0-6) after Week 0 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 60 | 59 | 58 | 60 | 60 | 59 | 60 | 59
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Any Irritability/Fussiness | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Any Loss of appetite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fever | 8 | 9 | 6 | 3 | 4 | 2 | 4 | 4

26. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: as for outcome 25
Time Frame: Within 7 days (Days 0-6) after Week 6 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 55 | 55 | 54 | 57 | 57 | 55 | 58 | 51
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Irritability/Fussiness | 1 | 1 | 6 | 1 | 3 | 3 | 0 | 2
  Any Loss of appetite | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Any Fever | 6 | 9 | 10 | 4 | 10 | 7 | 7 | 9

27. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: as for outcome 25
Time Frame: Within 7 days (Days 0-6) after Week 10 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 52 | 54 | 51 | 54 | 56 | 51 | 57 | 51
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Irritability/Fussiness | 3 | 2 | 0 | 1 | 0 | 1 | 0 | 1
  Any Loss of appetite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fever | 11 | 7 | 6 | 6 | 4 | 7 | 2 | 2

28. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: as for outcome 25
Time Frame: Within 7 days (Days 0-6) after Week 14 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 51 | 53 | 51 | 54 | 55 | 50 | 57 | 52
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Irritability/Fussiness | 4 | 2 | 4 | 0 | 1 | 2 | 1 | 2
  Any Loss of appetite | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Fever | 9 | 5 | 10 | 2 | 2 | 10 | 3 | 4

29. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: Solicited general symptoms assessed include Drowsiness, Fever (temperature by axillary route ≥ 37.5°C), Irritability/Fussiness and Loss of appetite. "Any" about a specific symptom is defined as incidence of this symptom, regardless of its intensity or relationship to vaccination. RTS,S Neo-10-14 Group, RTS,S 6-10-14 Group and Engerix-B Neo Group didn't receive any vaccination at this time point
Time Frame: Within 7 days (Days 0-6) after Week 26 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-26 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group
Number analyzed (Participants) | 49 | 54 | 54 | 46 | 56
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 | 0
  Any Irritability/Fussiness | 0 | 0 | 0 | 2 | 2
  Any Loss of appetite | 0 | 0 | 0 | 0 | 1
  Any Fever | 8 | 7 | 2 | 7 | 10

30. Secondary Outcome: Number of Subjects Reported With Solicited General Symptoms
Description: as for outcome 25
Time Frame: Within 7 days (Days 0-6) after Month 9 vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 50 | 49 | 48 | 54 | 51 | 47 | 56 | 51
Participants
  Any Drowsiness | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Any Irritability/Fussiness | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0
  Any Loss of appetite | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  Any Fever | 1 | 5 | 6 | 2 | 3 | 2 | 10 | 1

31. Other Pre Specified Outcome: Concentrations of Antibodies Against Circumsporozoite Protein of Plasmodium Falciparum (Anti-CS Antibodies)
Description: Month 18 immunogenicity data were tertiary objectives, and although not required to be disclosed were included in this result summary at the request of the study team to show the full study immunogenicity results.
Time Frame: At Month 18 post vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 45 | 43 | 47 | 47 | 45 | 40 | 52 | 48
EL.U/mL | 5.1 [3.1 to 8.3] | 12.7 [7.2 to 22.3] | 12 [8.3 to 17.4] | 16.2 [9.4 to 28.1] | 14.3 [8.7 to 23.6] | 33.8 [24.7 to 46.4] | 49.3 [36.2 to 67] | 0.3 [0.2 to 0.3]

32. Other Pre Specified Outcome: Anti-Hepatitis B Surface Antibody (Anti-HBs) Concentrations
Description: as for outcome 31
Time Frame: At Month 18 post vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
Number analyzed (Participants) | 40 | 41 | 45 | 45 | 43 | 39 | 47 | 42
mIU/mL | 1656.6 [1180.1 to 2325.4] | 3509.9 [2464.8 to 4998] | 1823.1 [1260.6 to 2636.5] | 4208.4 [3045.5 to 5815.5] | 4725.7 [3508.7 to 6364.7] | 7341.5 [5023.1 to 10729.9] | 12045.3 [8881.5 to 16336.2] | 78 [44.1 to 137.9]

ADVERSE EVENTS:
Time Frame: Solicited symptoms: Within 7 days (Days 0-6) after vaccination at Weeks 0, 6, 10, 14, 26 and Month 9; SAES: During the entire study period, from Month 0 to Month 18 (corresponding data lock point date = 23 March 2015)
Description: Unsolicited AEs: During the 30-day (Days 0-29) post vaccination period following 3 doses of RTS,S/AS01E versus DTPwHepB/Hib for the Engerix-B Neo Group. Please note that safety analysis for solicited symptoms and unsolicited AEs was performed only on subjects with available results.
Arm/Group | RTS,S Neo-10-14 Group | RTS,S Neo-10-26 Group | RTS,S 6-10-14 Group | RTS,S 6-10-26 Group | Engerix-B Neo/RTS,S 6-10-26 Group | RTS,S 10-14-26 Group | RTS,S 14-26-9M Group | Engerix-B Neo Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/59 | 0/60 | 0/60 | 0/60 | 1/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 7/60 | 5/59 | 6/60 | 9/60 | 8/60 | 12/60 | 5/60 | 4/60
Other Adverse Events (participants affected / at risk) | 36/60 | 35/59 | 28/58 | 29/60 | 35/60 | 36/59 | 47/60 | 31/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTS,S Neo-10-14 Group (N=60) | RTS,S Neo-10-26 Group (N=59) | RTS,S 6-10-14 Group (N=60) | RTS,S 6-10-26 Group (N=60) | Engerix-B Neo/RTS,S 6-10-26 Group (N=60) | RTS,S 10-14-26 Group (N=60) | RTS,S 14-26-9M Group (N=60) | Engerix-B Neo Group (N=60)
Gastroenteritis (Infections and infestations) | 4 | 0 | 2 | 2 | 4 | 5 | 2 | 1
Bronchiolitis (Infections and infestations) | 2 | 3 | 1 | 2 | 2 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 2 | 1 | 1 | 3 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drowning (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis neonatal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | RTS,S Neo-10-14 Group (N=60) | RTS,S Neo-10-26 Group (N=59) | RTS,S 6-10-14 Group (N=58) | RTS,S 6-10-26 Group (N=60) | Engerix-B Neo/RTS,S 6-10-26 Group (N=60) | RTS,S 10-14-26 Group (N=59) | RTS,S 14-26-9M Group (N=60) | Engerix-B Neo Group (N=59)
Pyrexia (General disorders) | 3 | 2 | 5/54 | 1/57 | 5/57 | 2/52 | 3/57 | 1/52
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3/54 | 2/57 | 3/57 | 1/52 | 2/57 | 2/52
Bronchiolitis (Infections and infestations) | 0 | 0 | 1/54 | 3/57 | 2/57 | 0/52 | 0/57 | 0/52
Conjunctivitis (Infections and infestations) | 4 | 5 | 1/54 | 2/57 | 2/57 | 6/52 | 5/57 | 2/52
Gastroenteritis (Infections and infestations) | 3 | 5 | 0/54 | 3/57 | 2/57 | 9/52 | 8/57 | 2/52
Malaria (Infections and infestations) | 5 | 3 | 2/54 | 0/57 | 4/57 | 5/52 | 9/57 | 0/52
Nasopharyngitis (Infections and infestations) | 6 | 3 | 6/54 | 6/57 | 3/57 | 3/52 | 7/57 | 7/52
Oral candidiasis (Infections and infestations) | 1 | 3 | 0/54 | 0/57 | 1/57 | 1/52 | 1/57 | 0/52
Pneumonia (Infections and infestations) | 8 | 6 | 3/54 | 7/57 | 6/57 | 5/52 | 9/57 | 6/52
Respiratory tract infection (Infections and infestations) | 1 | 2 | 0/54 | 3/57 | 1/57 | 0/52 | 1/57 | 0/52
Upper respiratory tract infection (Infections and infestations) | 11 | 15 | 10/54 | 6/57 | 11/57 | 13/52 | 15/57 | 13/52
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3/54 | 0/57 | 5/57 | 2/52 | 4/57 | 3/52
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 0/54 | 2/57 | 3/57 | 5/52 | 2/57 | 2/52
Pain (General disorders) | 4 | 5 | 7 | 7 | 4 | 6 | 5 | 6
Redness (General disorders) | 4 | 5 | 6 | 6 | 7 | 5 | 11 | 6
Swelling (General disorders) | 7 | 5 | 6 | 8 | 6 | 6 | 8 | 6
Irritability (General disorders) | 4 | 2 | 6 | 1 | 3 | 3 | 1 | 2
Fever (axillary temperature >= 37.5°C) (General disorders) | 11 | 9 | 10 | 6 | 10 | 10 | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.